CLINICAL TRIAL: NCT02458521
Title: A Study of Bilateral Prefrontal Transcranial Magnetic Stimulation (TMS) to Treat the Symptoms of Mild TBI (mTBI) and PTSD
Brief Title: Transcranial Magnetic Stimulation (TMS) to Treat mTBI and PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol # [397662]; CNRM 0048 (Other: Center for Neuroscience and Regenerative Medicine (CNRM))
Record Dates: First submitted 2015-04-30; First posted 2015-06-01 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Traumatic Brain Injury; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Magnetic Stimulation (Experimental): TMS sessions will consist of both 10Hz left pre-frontal stimulation for 3,500 pulses followed by 1Hz right pre-frontal stimulation for 1,500 pulses per session, for a total stimulation time of approximately one hour per session.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham TMS treatments will be conducted five times a week for 5 consecutive weeks, followed by a tapering of three sessions during week 6 and two sessions during week 7.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Treatment will consist of 30 sessions of TMS over approximately 7 weeks. More specifically, the active or sham TMS treatments will be conducted five times a week for 5 consecutive weeks, followed by a tapering of three sessions during week 6 and two sessions during week 7. TMS sessions will consist of both 10 Hz left pre-frontal stimulation for 3,500 pulses followed by 1 Hz right pre-frontal stimulation for 1,500 pulses per session, for a total stimulation time of approximately one hour per session. These pulse sequences have theoretical targets that may be implicated in conditions of poor resiliency, apathy, depression and anxiety.
  Arms: Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — Treatment will consist of 30 sessions of TMS over approximately 7 weeks. More specifically, the active or sham TMS treatments will be conducted five times a week for 5 consecutive weeks, followed by a tapering of three sessions during week 6 and two sessions during week 7. The TMS system will have three coils, one designated active and the other two unlabeled and identical in appearance, weight, and noises emitted, one of which will be active and one of which will be sham.
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
The overall objective of this project is to determine the efficacy and tolerability of TMS for mild Traumatic Brain Injury (mTBI) with PTSD symptoms and correlate treatment response with anatomical and biological factors unique to each service member (SM). Exploratory work will be done to look at the neuronal and biological changes that may occur over the course of TMS treatment.

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. To assess the change on the Rivermead Post-Concussion Symptoms Questionnaire (RPQ) and the PTSD Check List-Civilian Version (PCL-C) administered pre-treatment, then bi-weekly (weeks 2, 4, 6) during a 7 week treatment course, then monthly for 3 months following treatment.

   Hypothesis: The addition of high frequency left pre-frontal and low frequency right pre-frontal cortical stimulation will improve symptom reporting on the RPQ and PCL-C in service members with mTBI and PTSD symptoms as compared to sham treatment.
2. To assess the tolerability of TMS in subjects as measured by side effects in active TMS compared with sham treatment.

Hypothesis: TMS will prove safe and tolerable in service members with mTBI and PTSD.

The secondary objectives of this study are:

1. To assess whether TMS results in an improvement in mood as measured by the Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR), general life functioning (physical, cognitive, emotional, behavioral, and social problems) as measured by the Mayo-Portland Adaptability Inventory - military (MPAI-m), life satisfaction as measured by the Satisfaction With Life Scale (SWLS), and suicidality as measured by the Beck Scale for Suicidal Ideation (BSS).

   Hypothesis: TMS will result in an improvement in mood, general life functioning, and life satisfaction, as well as a reduction in suicidality.
2. To assess the durability of any improvement realized by TMS over the course of three months following the conclusion of sessions.

   Hypothesis: The improvement realized by 7 weeks of TMS will prove stable, showing effects up to 3 months after the conclusion of active treatment.
3. To assess structural neuronal changes over the course of active vs. sham TMS as measured by MRI.

   Hypothesis 1: Analysis of structural MRI (3D T1-weighted) will reveal increased volume of the hippocampus and anterior cingulate cortex in service members who improve in PTSD symptoms (as measured by the PCL-C).

   Hypothesis 2: Microstructural MRI (DTI) will reveal FA increase in the corpus callosum and the uncinated fasciculus in service members who improve in measures of mTBI (i.e., Rivermead Post Concussion Symptoms Questionnaire).
4. To assess metabolic neuronal changes that occur over the course of active vs. sham TMS as measured by PET.

   Hypothesis 1: TMS will result in increased glucose uptake in the ipsilateral and contralateral cerebral hemispheres for those who show significant improvements in the symptomatic measures of TBI (i.e. RPQ and MPAI-m).

   Hypothesis 2: TMS will result in decreased glucose uptake in the dorsal anterior cingulate/mid cingulate cortex (dACC/MCC) and in the bilateral amygdala for those service members with significant improvements in the symptomatic measures of PTSD and mood (i.e. PTSD Checklist and QIDS-SR).
5. To examine the mechanism of action of TMS through looking at the metabolic changes that occur during a TMS session.

   Hypothesis: There will be increased glucose uptake in the left prefrontal cortex and decreased glucose uptake in the right prefrontal cortex immediately after active TMS as compared to sham.
6. Exploratory: To assess biological changes that result from TMS therapy and to determine how biomarkers relate to changes in PTSD symptoms.
7. Exploratory: To examine how single gene polymorphisms (SNPs) in serotonin genes may relate to TMS response and symptom change.

ELIGIBILITY:
Inclusion Criteria:

1. Military health care beneficiary for enrollment (loss of benefits will not require separation from the study).
2. Over the age of 18 years.
3. Presence of mTBI (based on standard Veterans Affairs (VA)/ Department of Defense (DoD) criteria).
4. Presence of PTSD symptoms (PCL score over 30).

Exclusion Criteria:

1. Evidence of moderate or severe TBI (based on standard VA/DoD criteria). Incidental neuroimaging findings that may or may not be related to trauma (e.g. white matter hyperintensities on structural MRI) are not sufficient to identify a subject as a moderate TBI if other severity markers fall in the mild TBI range.
2. History of seizure, bipolar disorder, schizophrenia, or current dependence to psychoactive substance(s).
3. History of severe or recent heart disease.
4. Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain.
5. Use of medications that potentially lower seizure threshold without concomitant administration of anticonvulsant drugs which may protect against seizure occurrence.
6. Not a suitable candidate for the study as determined by the PI.
7. Pregnancy or plans to become pregnant during the course of the study (determined via urine-pregnancy test).
8. Presence of metallic hardware in close contact to the discharging coil (e.g. cochlear implants, internal pulse generator).
9. Presence of implanted brain electrodes (cortical or deep-brain electrodes).
10. MRI portion: Presence of metal fragments or devices (cardiac pacemaker, neural stimulator, etc.), which are determined by a radiologist to contraindicate MRI (at 3 Tesla). Also, presence of metal (such as dental braces) which causes significant degradation of the MRI signal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Rivermead Post-Concussion Symptoms Questionnaire (RPQ) | Measured to compare changes from Baseline; during weeks 2, 4, and 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.
  The RPQ gauges the severity of post-concussion symptoms. The subject rates thMeasured to compare changes from Baseline; during weeks 2, 4, 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.e degree to which 16 symptoms are more of a problem compared with premorbid levels from 0 (not experienced at all) to 4 (a severe problem). The questionnaire has been shown to have good test-retest reliability.
PTSD Check List-Civilian (PCL-C) | Measured to compare changes from Baseline; during weeks 2, 4, and 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.
  The PCL-C is a self-report questionnaire on the presence and severity of PTSD symptoms. The questionnaire asks subjects how much they are affected by each of 17 PTSD symptoms in the last month on a scale ranging from 1 (not at all) to 5 (extremely) to yield a total PTSD symptom severity score and subscale scores on (a) re-experiencing (b) avoidance (c) arousal. The PCL-C has been shown to demonstrate excellent internal consistency and convergent validity with other measures of PTSD.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) | Measured to compare changes from Baseline; during weeks 2, 4, 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.
  QIDS-SR is a shortened version of the Inventory of Depressive Symptomatology, Self-report (IDS-SR) that covers just items that assess DSM-IV criterion diagnostic symptoms for depression. The QIDS-SR contains 16 items that separate into the nine DSM-IV symptom domains of (1) sadness (2) concentration (3) self-criticism (4) suicidal ideation (5) interest (6) energy/fatigue (7) sleep disturbance (8) decrease/increase in appetite/weight and (9) psychomotor agitation/retardation. Research indicates that the IDS-SR has high internal consistency and shows convergent validity with the IDS-SR and the Hamilton Rating Scale for Depression (HAM-D).
Beck Scale for Suicide Ideation (BSS) | Measured to compare changes from Baseline; during weeks 2, 4, 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.
  The BSS is a measure that quantifies the intensity of current conscious suicidal intent by scaling various dimensions of self-destructive thoughts or desires. The BSS has been shown to have high internal consistency, construct validity, and be sensitive to changes in depression and hopelessness.
Mayo-Portland Adaptability Inventory-Military Edition (MPAI-m) | Measured to compare changes from Baseline; during weeks 2, 4, 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.
  The MPAI-m is a modified version of the Mayo-Portland Adaptability Inventory-Fourth Edition (MPAI-4), which has been shown to have internal consistency, construct validity, predictive validity, sensitivity to treatment effects, and have convergent validity with the Disability Rating Scale and the Rancho Scale. The MPAI-m is a reliable measure that shows satisfactory construct validity in the assessment of functional abilities and activity in military members with mild TBI.
Satisfaction with Life Scale (SWLS) | Measured to compare changes from Baseline; during weeks 2, 4, 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.
  The SWLS is designed to measure satisfaction with life as a whole. The measure consists of marking agreement on a scale from 1 (strongly disagree) to 7 (strongly agree) on five items pertaining to general life satisfaction. The SWLS has been shown to possess good convergent validity with other scales and assessments of subjective well-being, temporal stability, sensitivity to changes in life satisfaction over the course of clinical intervention, and discriminant validity from emotional well-being measures.

OTHER OUTCOMES:
Pain Rating | Measured to compare changes from Baseline; during weeks 2, 4, 6 of treatment; and during the Month 1, Month 2, and Month 3 follow up visits after treatment ends.
  Subjects will be assessed for potential pain syndromes prior to undergoing active or sham TMS. If one or more pain syndromes are present, data will be collected regarding pain location, quality, and intensity as measured by a visual analogue scale (VAS) in terms of (1) average pain over the past week and (2) the worst incident of pain over the past week. The VAS is a simple and efficient minimally intrusive measure of pain, which has been widely used in clinical and research settings. The VAS has been experimentally examined and has been found to be a valid, internally consistent and reliable measure of pain. Subjects will be queried as to whether they have experienced pain (in terms of location, quality, and intensity as measured by VAS) during, or immediately after, the TMS procedure after each application of active or sham TMS.
Automated Neuropsychological Assessment Metrics (ANAM) | Will be administered 3 times to compare changes from (1) Baseline (within 30 days of initiating TMS or Sham treatment); (2) prior to a session during week 2 of TMS or Sham treatment; and (3) at the completion of TMS or Sham treatment (week 7).
  The Automated Neuropsychological Assessment Metrics (ANAM) is a library of computer-based 22 assessments that are sensitive to cognitive change in attention, concentration, the standard neurocognitive assessment employed by all services in the Department of Defense. The ANAM takes approximately 20 minutes to administer.
Structural Neuronal Changes to be assessed by MRI Assessment | Measured at Baseline and compared to results at completion of treatment (week 7).
  Neurologic MR imaging will be on a 3.0 Tesla MR Scanner equipped with a high-performance gradient subsystem. MRI will be performed at the NICoE with data analysis and storage by the Image Processing Core of the Center for Neuroscience and Regenerative Medicine (CNRM).
  The MRI testing will utilize the standard NICoE TBI scan suite. Currently, this may include Hi-resolution T1 and T2 anatomic scans, FLAIR, DTI, fMRI, and Gd-perfusion. Scan sequences for all subjects will be as similar as possible. Total scan duration will not exceed 90 minutes.
Metabolic Neuronal Changes to be assessed by PET Assessment (FDG-PET) | Measured at Baseline and compared to results from week 2 of treatment, and at completion of treatment (week 7).
  Following a minimum 4-hour fasting period, a finger stick blood glucose level is performed. An intravenous dose of 5 millicuries (mCi) FDG is then administered followed by quiet resting in the supine position in a darkened room for 50 (+/- 5) minutes. Co-registered (fusion) low dose computed axial tomographic (CT) images followed by positron emission tomographic (PET) images of the brain are then obtained on a PET-CT scanner (Siemens Biograph mCT, Siemens Medical Solutions).
  In the case of the second PET, the subject will be injected with the FDG immediately prior to undergoing a single TMS or Sham treatment session and will then obtain the CT and PET imaging post completion of the active or sham TMS session. This will allow the investigational team to examine correlations between symptom treatment response and areas within the brain that demonstrated either activation or inhibition during TMS treatment as measured through PET.
Biomarker Assessment: Blood Samples | Measured at Baseline and compared to changes at week 7 of treatment, and the Month 3 follow-up visit post-treatment.
  Samples will be each assigned a unique identifying code to ensure patient privacy and will be processed and maintained within the CNRM repository following all IRB and regulatory requirements.
  Upon collection, biomarkers will be sent to the CNRM Biospecimen Repository, located in Rockville, Maryland for storage.
Biomarker Assessment: Saliva Samples | Measured at Baseline and compared to changes at week 7 of treatment, and the Month 3 follow-up visit post-treatment.
  Samples will be each assigned a unique identifying code to ensure patient privacy and will be processed and maintained within the CNRM repository following all IRB and regulatory requirements.
  Upon collection, biomarkers will be sent to the CNRM Biospecimen Repository, located in Rockville, Maryland for storage.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey G Grammer, M.C., Study Chair — National Intrepid Center of Excellence; Paul F Pasquina, M.D., Principal Investigator — Walter Reed National Military Medical Center; Louis M French, Psy.D, Study Chair — Walter Reed National Military Medical Center; Nancy de Almeida, RN, Study Chair — Walter Reed National Military Medical Center
Locations (1):
- National Intrepid Center of Excellence, Walter Reed National Military Medical Center, Bethesda, Maryland, United States